CLINICAL TRIAL: NCT04795570
Title: Hormonal Status and Coagulative Disorders as Risk Factors for Urethral Stricture After Transurethral Resection of the Prostate/Bladder: A Prospective Study
Brief Title: Urethral Stricture After Transurethral Resection of the Prostate/Bladder: a Prospective Study of Risk Factors
Acronym: STRICT-TURP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Virgen de las Nieves (Other)
Collaborators: Instituto de Investigación Biosanitaria de Granada (ibs.Granada) (Unknown)
Responsible Party: Principal Investigator, Ignacio Puche Sanz, MD PhD, University Hospital Virgen de las Nieves
Other Study IDs: RTU_EstenosisUretra_2020_HUVN
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Urethral Stricture, Male; Hormone Deficiency; Fibrosis
MeSH Terms: conditions — Urethral Stricture; Fibrosis | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases. Patients who develop urethral stricture: Patients who develop urethral stricture within 6 months after TUR P/B
  Interventions: Procedure: Transurethral resection of the prostate or bladder
- Controls. Patients who DO NOT develop urethral stricture: Patients who DO NOT develop urethral stricture within 6 months after TUR P/B
  Interventions: Procedure: Transurethral resection of the prostate or bladder

INTERVENTIONS:
Procedure: Transurethral resection of the prostate or bladder — All patients undergoing TUR P/B will undergo a blood draw within 6 months after surgery to determine hormonal status and coagulation disorders.

SUMMARY:
There is currently no prognostic or predictive risk marker for this urethral stricture disease.

The most conservative standard treatment for urethral stricture (internal urethrotomy) has a very high recurrence rate (greater than 75%) and, on many occasions, reconstructive urologists have to choose within a great variety of further complex interventions. Knowing risk and predictive markers of this disease could help to optimize both the need and the approach for these surgeries and may offer a more individualized management to patients.

DETAILED DESCRIPTION:
The pathophysiological mechanisms that influence the development of urethral stricture are not established. In developed countries, the most common etiology of urethral stricture is idiopathic (41%) followed by iatrogenic (35%).

Serum testosterone is important in urethral development, in the integrity of the corpora cavernosa and has been shown to play a fundamental role in the development of genital structures. Recently, hypoandrogenism (HA) has been associated with a decrease in urethral androgen receptors and periurethral vascularization. Furthermore, low serum testosterone levels appear to be implicated in an increased risk of urethral atrophy.

In recent years it has been proven that coagulation, in addition to influencing the formation of the provisional matrix, participates in mechanisms of tissue injury through the activation of PARs. As a result, the coagulation cascade directly influences several key aspects of the wound healing response, from platelet aggregation and vasoconstriction, but also inflammation and scar formation. Although it is strictly regulated under normal conditions, an imbalance in favor of a procoagulant state as occurs in many pathologies of other organs (liver, lung, kidney) has the potential to deregulate inflammatory and tissue repair mechanisms and culminate in fibrosis.

In general, it is accepted that the probability of developing a urethral stricture after endoscopic treatment is around 2-10% of cases. However, this complication has never been studied in depth and the true incidence of urethral stricture, and its consequences in quality of life, after a transurethral procedure is unknown.

The aim of this study is to analyze the potential role of serum hormonal status and coagulation disorders as risk factors for the development of urethral stricture after transurethral surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing transurethral resection of the prostate or bladder (TUR P/B) at our department.

Exclusion Criteria:

* Patients not giving their informed consent
* Patients with urethral catheter at the moment of TUR P/B
* Patients with any type of urethral stricture at the moment of TUR P/B
* Patients under hormonal treatments (testosterone, thyroxine...) 1 year before the TUR P/B.
* Patients with already known coagulation disorders or undergoing anticoagulation treatments at the moment of the blood test.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing transurethral resection of the prostate or bladder
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Development of anatomic urethral stricture | 6 months
  It will be studied in all patients by flexible urethroscopy

SECONDARY OUTCOMES:
Development of functional urethral stricture | 6 months
  Studied by uroflowmetry and PROM questionnaries

OTHER OUTCOMES:
Hormonal status | Within 6 months after TUR P/B
  Determination of serum sexual hormones (Testosterone, estrogens, FSH, LH), TSH, T4 and PRL
Coagulation disorders | The day before TUR P/B
  Comprehensive profile of procoagulation disorders determined in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Puche-Sanz, MD PhD, Principal Investigator — University Hospital Virgen de las Nieves
Locations (1):
- Hospital Universitario Virgen de las Nieves, Granada, Spain

IPD SHARING:
Plan to Share IPD: No